CLINICAL TRIAL: NCT07345728
Title: A Clinical Study Evaluating the Safety and Efficacy of BAFFR CAR-T Therapy for Relapsed/Refractory B-cell Malignancies
Brief Title: Clinical Study Evaluating the Safety and Efficacy of BAFFR CAR-T Therapy for Relapsed/Refractory B-cell Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Donghua Zhang (Other)
Responsible Party: Sponsor-Investigator, Donghua Zhang, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHZ1962-A
Record Dates: First submitted 2025-12-16; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory B-cell Malignancies
Keywords: relapsed/refractory B-cell malignancies
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental:Experimental group (Experimental)
  Interventions: Drug: Infusion of BAFFR CAR-T therapy for relapsed/refractory B-cell malignancies

INTERVENTIONS:
Drug: Infusion of BAFFR CAR-T therapy for relapsed/refractory B-cell malignancies — Infusion of BAFFR CAR-T therapy for relapsed/refractory B-cell malignancies

SUMMARY:
This is a prospective, single-arm, multi-center, randomized controlled clinical study designed to evaluate the safety and efficacy of BAFFR CAR-T therapy for relapsed/refractory B-cell malignancies. A total of 30 subjects are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Patients or their guardians understand and voluntarily sign the informed consent form, and are expected to complete the follow-up examinations and treatment procedures of the study; Age 18-85 years (inclusive), gender not restricted; Patients with relapsed/refractory B-cell lymphoma who have received prior treatment including anti-CD20 targeted agents (unless documented CD20 negative) and anthracycline-containing regimens; Pathological immunohistochemistry of tumor confirms positive BAFFR target expression at screening; Patients have recovered from the toxicities of previous treatments, i.e., CTCAE toxicity grade < 2 (unless abnormalities are tumor-related or judged by the investigator to be stable and not significantly affecting safety or efficacy); ECOG performance status 0-2 and life expectancy > 3 months;

Adequate organ function:

1. Alanine transaminase (ALT) ≤ 3 × upper limit of normal (ULN);
2. Aspartate transaminase (AST) ≤ 3 × ULN;
3. Total bilirubin ≤ 1.5 × ULN;
4. Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 60 mL/min;
5. Hemoglobin ≥ 60 g/L or maintained at this level after transfusion;
6. Room air oxygen saturation ≥ 92%;
7. Left ventricular ejection fraction (LVEF) ≥ 45%; Accessible venous access for apheresis and no contraindications to leukapheresis.

Exclusion Criteria:History of other malignancies within 3 years prior to screening, except for adequately treated carcinoma in situ of the cervix, papillary thyroid cancer, basal or squamous cell skin cancer, localized prostate cancer after radical therapy, and ductal carcinoma in situ after radical therapy; Positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA titer above the lower limit of detection of the research institution; positive for hepatitis C virus (HCV) antibody with positive peripheral blood HCV-RNA; positive for human immunodeficiency virus (HIV) antibody; History of severe allergies [severe allergy is defined as grade 2 or higher allergic reaction with any of the following clinical manifestations: airway obstruction (runny nose, cough, wheezing, dyspnea), tachycardia, hypotension, arrhythmia, gastrointestinal symptoms (nausea, vomiting), incontinence, laryngeal edema, bronchospasm, cyanosis, shock, respiratory or cardiac arrest] or known hypersensitivity to any active ingredients, excipients, murine products, or xenogeneic proteins contained in this study (including lymphodepletion regimen); History of severe cardiac disease, including but not limited to severe arrhythmia, unstable angina, massive myocardial infarction, New York Heart Association class III or IV cardiac insufficiency, myocardial infarction or coronary artery bypass grafting (CABG) within ≤ 6 months prior to screening, history of unexplained syncope not due to vasovagal reaction or dehydration, history of severe non-ischemic cardiomyopathy, refractory hypertension (refractory hypertension is defined as: despite lifestyle modifications, blood pressure remains uncontrolled after > 1 month of treatment with reasonable, tolerable, and adequate doses of ≥ 3 antihypertensive drugs (including diuretics), or requires ≥ 4 antihypertensive drugs to achieve effective blood pressure control); Unstable systemic disease as judged by the investigator: including but not limited to severe liver, kidney, or metabolic diseases requiring medical treatment; Previous organ transplantation or planned organ transplantation (except hematopoietic stem cell transplantation); Active autoimmune or inflammatory neurological diseases (e.g., Guillain-Barré syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular disease (e.g., cerebral edema, posterior reversible encephalopathy syndrome (PRES)); Presence of tumor emergencies (e.g., spinal cord compression, bowel obstruction, leukostasis, tumor lysis syndrome, etc.) requiring urgent treatment at screening or before infusion; Uncontrolled bacterial, fungal, viral, or other infections requiring antibiotic treatment; Use of short-acting hematopoietic growth factors affecting blood counts within 1 week, or long-acting hematopoietic growth factors within 2 weeks prior to planned CAR-T manufacturing apheresis, and judged by the investigator to affect cell manufacturing;

Receiving corticosteroids or immunosuppressive drugs within 2 weeks prior to planned CAR-T manufacturing apheresis, and judged by the investigator to affect cell manufacturing:

1. Corticosteroids: Subjects receiving systemic steroid therapy within 2 weeks prior to planned CAR-T manufacturing apheresis and judged by the investigator to require long-term systemic steroid therapy during treatment (except inhaled or topical use); and subjects receiving systemic steroid therapy within 72 hours before cell infusion (except inhaled or topical use);
2. Immunosuppressants: Subjects receiving immunosuppressive agents within 2 weeks prior to planned CAR-T manufacturing apheresis; Major surgery (except diagnostic procedures and biopsies) within 4 weeks prior to lymphodepletion or planned major surgery during the study, or incompletely healed surgical wounds before enrollment; Vaccination with (live-attenuated) viral vaccines within 4 weeks prior to screening; History of severe mental illness; History of alcoholism or substance abuse; Pregnant or lactating women, and female subjects planning pregnancy within 2 years after cell infusion or male subjects whose partners plan pregnancy within 2 years after their cell infusion; Subjects with contraindications to any study procedures or other medical conditions that may pose unacceptable risks according to the investigator's judgment and/or clinical standards.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 1,3,6,12,18,24 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, China